CLINICAL TRIAL: NCT01130714
Title: Effectiveness of a Resistance Training Program on Inflammatory Markers and Chemotherapy Completion in Lung Cancer Patients on Chemotherapy
Brief Title: Resistance Training in Lung Cancer Patients on Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Kristina Karvinen, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCIRB 09-0725
Record Dates: First submitted 2010-01-06; First posted 2010-05-26 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Inflammation; Lung Cancer
Keywords: inflammation; chemotherapy; lung cancer
MeSH Terms: conditions — Inflammation; Lung Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training (Experimental): Group assigned to complete resistance training during duration of chemotherapy.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Exercise — Resistance training with resistance bands.
  Arms: Resistance training

SUMMARY:
The purpose of this study is to examine the effectiveness of a resistance training program on reducing systemic inflammation and improving chemotherapy completion in lung cancer patients being treated with curative intent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed with lung cancer
* Stage I, II, or III
* Eligible for chemotherapy with curative intent
* 21 years of age or older
* Approval to participate in study by treating oncologist or family physician

Exclusion Criteria:

* Unstable cardiac disease
* Untreated bone or brain metastases

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Systemic inflammation measured by c-reactive protein. | 12 weeks

SECONDARY OUTCOMES:
Chemotherapy completion | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristina H Karvinen, PhD, Principal Investigator — East Carolina University
Locations (1):
- Leo Jenkins Cancer Center, Greenville, North Carolina, United States

REFERENCES:
- [Derived] Karvinen KH, Esposito D, Raedeke TD, Vick J, Walker PR. Effect of an exercise training intervention with resistance bands on blood cell counts during chemotherapy for lung cancer: a pilot randomized controlled trial. Springerplus. 2014 Jan 8;3:15. doi: 10.1186/2193-1801-3-15. eCollection 2014. PMID 24683529